CLINICAL TRIAL: NCT06329622
Title: Ketosteril Sarcopenia Chronic Kidney Disease
Brief Title: Effect of Ketosteril on Sarcopenia in Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chen Jing, Director of Nephrology, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-972
Record Dates: First submitted 2023-11-17; First posted 2024-03-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease; Sarcopenia
Keywords: CKD; sarcopenia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia | interventions — Diet, Protein-Restricted; ketosteril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the intervention group, low-protein diet (0.6-0.8g protein/kg body weight/day) and Ketosteril 0.12 g/kg body weight/day will be prescribed with the target energy intake of 25-30kcal/kg body weight/day. The intervention will last for 6 months. Then,during the subsequent 3-month observation period, the patients maintain a low-protein diet (0.6-0.8g protein/kg body weight/day) with the target energy intake of 25-30kcal/kg body weight/day.
  Interventions: Combination Product: low-protein diet + Ketosteril
- Control (Active Comparator): In the control group, low-protein diet (0.6-0.8g protein/kg body weight/day) and the target energy intake of 25-30kcal/kg body weight/day will be prescribed for 9 months
  Interventions: Dietary Supplement: low-protein diet

INTERVENTIONS:
Combination Product: low-protein diet + Ketosteril — low-protein diet (0.6-0.8g protein/kg body weight/day) and Ketosteril 0.12 g/kg body weight/day will be prescribed with the target energy intake of 25-30kcal/kg body weight/day.
  Arms: Intervention
Dietary Supplement: low-protein diet — low-protein diet (0.6-0.8g protein/kg body weight/day) with the target energy intake of 25-30kcal/kg body weight/day.
  Arms: Control

SUMMARY:
The investigators hypothesize that Ketosteril can improve sarcopenia in patients with renal disease without increasing the burden on the kidneys and causing deterioration of renal function. Therefore, this study intends to take patients with CKD stage 3-4 and sarcopenia as the research object, give Ketosteril intervention or not to patients on the base of low-protein diet, and clarify the clinical benefits of Ketosteril prescription for improving sarcopenia in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for CKD stage 3-4 (15 ≤eGFR<60 ml/(min*1.73m2)) in the 2012 Kidney Disease Improving Global Outcomes (KDIGO) guideline.
2. Sarcopenia should be diagnosed According to the 2019 Asian Working Group for Sarcopenia (AWGS) diagnostic criteria for sarcopenia: ① Muscle strength: grip strength (< 28 kg for males, < 18 kg for females); ② Physical function: is assessed by walking speed over 6 m (< 1.0 m/s) or five-repetition sit-to-stand test (5STS) (≥ 12 s) or recommended short physical performance battery (SPPB) (≤ 9); ③ Artificial skeletal muscle (ASM) of extremities: Bioelectrical impedance analyzer (BIA) (< 7.0 kg/m2 for males and < 5.7 kg/m2 for females). On the basis of meeting criteria ③, sarcopenia can be diagnosed if at least one of the first two items is met.
3. Patient can walk normally.
4. Provide the written informed consent.

Exclusion Criteria:

1. Patients with diabetes.
2. Obese/overweight patients (body mass index>25 kg/m2)
3. Had previously received renal replacement therapy (including kidney transplantation, hemodialysis, peritoneal dialysis).
4. Patients with new cardiovascular events, uncontrolled acute or chronic cardiac failure within 3 months.
5. Patients with acute infection (C-reactive protein>10 mg/L) or acute exacerbation of chronic diseases that is not under control within 3 months.
6. Patients with cerebrovascular events, severe liver disease, malignant tumor and multiple organ failure.
7. Patients with osteoarthritis, metabolic bone disease, osteonecrosis of the femoral head, hemiplegia and cognitive dysfunction.
8. Patients with hypercalcemia and amino acid metabolism disorder.
9. Those who are allergic to the active ingredients or other excipients of the Ketosteril.
10. Patients with poor compliance, unable to follow the study requirements for diet control.
11. Participated in other interventional clinical trials within 30 days before this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
skeletal muscle mass index (SMI) | six months after the intervention
  SMI=skeletal muscle weight/(height×height)，the muscle weight with the unit of kg and square of height with the unit of m2 will be combined to report SMI in kg/m^2

SECONDARY OUTCOMES:
changes in eGFR(ml/min/1.73m2) | six months after the intervention
  From baseline to the 6th month, changes in eGFR(ml/min/1.73m2)
serum albumin(g/l) | six months after the intervention
  From baseline to the 6th month, changes in serum albumin(g/l)
grip strength(kg) | six months after the intervention
  From baseline to the 6th month,changes in grip strength(kg)
BMI(kg/m2) | six months after the intervention
  From baseline to the 6th month,changes in BMI(kg/m2)
6m walking speed(s) | six months after the intervention
  From baseline to the 6th month,changes in 6m walking speed(s)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, PhD, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon request pending